CLINICAL TRIAL: NCT03051711
Title: An Open Label Study of GBT440 to Evaluate the Effect on Oxygenation in Healthy Subjects at Rest and Maximal Exercise Under Hypoxic Conditions
Brief Title: Study to Evaluate Effects of Investigational Drug on Oxygenation in Healthy Volunteers Under Hypoxic Conditions
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor discontinued IPF Program on 23-Oct. 2017 based on POC studies
Sponsor: Global Blood Therapeutics (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GBT440-0111
Expanded Access: NCT03943615 (No longer available)
Record Dates: First submitted 2017-01-18; First posted 2017-02-14 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Cardio-pulmonary Function
MeSH Terms: interventions — voxelotor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GBT440 Dose 1 (Experimental): Dose 1
  Interventions: Drug: GBT440
- GBT440 Dose 2 (Experimental): Dose 2
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — Capsules which contain GBT440 drug substance in Swedish Orange
  Other Names: 2-hydroxy-6-((2-(1-isopropyl-1H-pyrazol-5-yl)pyridin-3-yl)methoxy)benzaldehyde

SUMMARY:
To evaluate the effect of GBT440 on oxygen saturation at rest and exercise, under hypoxic conditions, at Day 15 compared to Baseline.

DETAILED DESCRIPTION:
This study in healthy subjects will evaluate GBT440 and its effects on cardio-pulmonary function under both normoxic and hypoxic conditions.

ELIGIBILITY:
INCLUSION CRITERIA

1. Males or females aged 18 - 50 years inclusive
2. Able and willing to provide signed informed consent to participate in this study
3. VO2 max ≥ 40 mL/kg/min for males, and ≥ 35 mL/kg/min for females
4. Weight ≥ 40 kg
5. Male or female of child bearing potential willing and able to use highly effective methods of contraception during the study to 30 days after the last dose of study drug.

EXCLUSION CRITERIA

1. Subjects whose exercise regimen at Screening is, in the Investigator's opinion, expected to change significantly during the study
2. Family or personal history of congenital long QT syndrome
3. Participated in another clinical trial of an investigational drug (or medical device) within 30 days or 5-half-lives, whichever is longer, prior to Screening, or is currently participating in another trial of an investigational drug (or medical device)
4. Clinically significant medical disease that is likely, in the Investigator's opinion, to significantly impact the study's efficacy and safety assessments (e.g., history significant cardio-pulmonary disease or arrhythmias) within 6 months of Screening.
5. AST, ALT or total bilirubin >2 × ULN
6. Serum creatinine >1.5 mg/dL
7. Clinical evidence of active infection, within 21 days of Screening, which may include but is not limited to bronchitis, pneumonia, urinary tract infection, or cellulitis.
8. Female who is breast-feeding or pregnant
9. Current smoker or history of smoking within 3 months from Screening
10. Any condition possibly affecting drug absorption, including but not limited to previous surgery on the stomach or small intestine
11. Known hypersensitivity to any component of the study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-12; Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
The change in oxygen saturation (%) at rest and exercise, under hypoxic conditions | Day 15

SECONDARY OUTCOMES:
Maximal oxygen uptake VO2 max (mL/kg/min) under normoxic and hypoxic conditions | Day 15
Cardiac output (L/min) under normoxic and hypoxic conditions | Day 15
Oxy-hemoglobin dissociation curve p50, under hypoxic conditions | Day 15
Perceived dyspnea score (1-10), under normoxic and hypoxic conditions | Day 15
Frequency and severity of treatment-emergent adverse events (TEAEs) as assessed by (NCI CTCAE Version 4.03) | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Balaratnam, MBChB, BAO, Study Director — Global Blood Therapeutics
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No